CLINICAL TRIAL: NCT00243893
Title: Tetracycline-Derivatives for Treatment of Cerebral Arteriovenous Malformations and Aneurysms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS027713 (NIH); NS034949; NCT00305994 (obsolete NCT alias)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Aneurysms; Arteriovenous Malformations
Keywords: giant aneurysms; arteriovenous malformations; minocycline; doxycycline; BAVM
MeSH Terms: conditions — Aneurysm; Arteriovenous Malformations; cyclopia sequence | interventions — Minocycline; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brain AVMs (Active Comparator): This trial is to investigate the use of minocycline or doxycycline as medical therapy, can minocycline or doxycycline induce biologically significant changes in the enzyme system thought to be related to spontaneous growth/rupture of these malformations. Finally, can patients safely tolerate these medications over an extended period of time.
  Interventions: Drug: minocycline; Drug: doxycycline
- Aneurysms (Active Comparator)
  Interventions: Drug: minocycline; Drug: doxycycline

INTERVENTIONS:
Drug: minocycline — Take minocycline 50mg BID x2 years. Labs drawn at baseline, then every-6 months. MRI is done at baseline and completion of study.
Drug: doxycycline — Take doxycycline 50mg BID x2 years. Labs drawn at baseline, then every-6 months. MRI is done at baseline and completion of study.

SUMMARY:
The purpose of this pilot study is to investigate the use of minocycline and doxycycline as medical therapy for inoperable or partially treated arteriovenous malformations (AVMs) and giant aneurysms.

DETAILED DESCRIPTION:
Arteriovenous malformations (AVMs) are a treatable cause of stroke in young adults. The processes by which AVMs and giant aneurysms grow in size and spontaneously bleed are unknown. The primary reason to treat AVMs and aneurysms is to guard against intracranial bleeding.

This pilot study will examine the use of two common antibiotics-minocycline and doxycycline-as medical therapy for inoperable or partially treated AVMs and giant aneurysms. These drugs, which are tetracycline derivatives, can reduce the levels of a family of enzymes, called matrix metalloproteases, that degrade tissue and thereby cause a reduction in the risk of spontaneous bleeding from AVMs or aneurysm-which is the main cause of stroke associated with these disorders. The enzymes can contribute to weaknesses in the wall of blood vessels and may increase the risk of the vessel wall rupturing and causing spontaneous bleeding.

This trial also will show that taking minocycline and doxycycline over an extended period in this patient population is safe and well tolerated. Results from this study could help plan future studies to benefit patients with abnormal blood vessels prone to bleeding in their brains.

ELIGIBILITY:
Inclusion Criteria:

* Giant aneurysms or brain arteriovenous malformations (BAVM)
* Female patients of child bearing age using effective birth control, males
* Creatinine no greater than 2.0 mg/dl
* ALT no greater than 2 times upper limit of control

Exclusion Criteria:

* Unstable medical illness
* Contraindications to Tetracycline
* History of vestibular disease, (except benign positional vertigo)
* Prior tetracycline use within 2 mos of baseline visit.
* History of noncompliance with treatment or other protocols
* History of systemic lupus
* Patients not eligible for MRI

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
MRI will be done baseline and post treatment. | 2 years
MMP levels are being followed q 6-mos. | Patients called weekly for 1st-3 months, then every 6-months until completion of study
Drug levels are being followed q 6-mos. | Patients called weekly for 1st-3 months, then every 6-months until completion of study

CONTACTS AND LOCATIONS:
Overall Officials: William L. Young, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

REFERENCES:
- [Result] Frenzel T, Lee CZ, Kim H, Quinnine NJ, Hashimoto T, Lawton MT, Guglielmo BJ, McCulloch CE, Young WL. Feasibility of minocycline and doxycycline use as potential vasculostatic therapy for brain vascular malformations: pilot study of adverse events and tolerance. Cerebrovasc Dis. 2008;25(1-2):157-63. doi: 10.1159/000113733. Epub 2008 Jan 23. PMID 18212521
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2605012/